CLINICAL TRIAL: NCT05148429
Title: Prenatal Screening of Intestinal Malrotation With a Higher Risk of Volvulus: Value of the Ultrasound Study of the Relative Position of the Superior Mesenteric Vessels and Fetal Abdominal MRI.
Brief Title: Prenatal Screening of Intestinal Malrotation With a Higher Risk of Volvulus.
Acronym: MALROT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0684
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Postnatal Complication; Mesenteric Pregnancy
Keywords: Pregnant women; 2nd trimester ultrasound examination; Mesenteric vessels positionning; Pediatric follow up +/- treatment; Postnatal confirmation; Evolution and complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fetuses with abnormal positionning of mesenteric vessels: All pregnant women with abnormal positionning of mesenteric vessels during second trimester scan
  Interventions: Other: Ultrasound exam; Other: Fetal MRI; Other: Postnatal abdominal ultrasound; Other: Pediatric Follow up

INTERVENTIONS:
Other: Ultrasound exam — Ultrasound exam
Other: Fetal MRI — Fetal MRI
Other: Postnatal abdominal ultrasound — Postnatal abdominal ultrasound
Other: Pediatric Follow up — Pediatric Follow up

SUMMARY:
Digestive malrotation is an anatomical anomaly of the positionning of the mesenteric vessels and the digestive tract that can lead in some form to a dangerous neonatal complication: intestinal volvulus. This requires emergency surgery with a risk of digestive resection. Visualizing during pregnancy the normal or abnormal anatomical positionning of the mesenteric vessels could make it possible to diagnose this malrotation and prevent the occurrence of this complication.

The aim of the study is to study the neonatal outcome of fetus confirm to have an abnormal positionning of mesenteric vessels

ELIGIBILITY:
Inclusion criteria:

* Pregnant women attending for 2nd trimester ultrasound
* Abnormal positionning of mesenteric vessels
* No other foetal malformation
* Singleton pregnancy
* Age >18 years

Exclusion criteria:

* Chromosomal abnormality
* polymalformative syndrom
* Foetal malformation changing intestine disposition (gastroschisis, diaphragmatic hernia, heterotaxis…)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women attending for 2nd trimester scan
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage of intestinal malrotation among foetuses | day 1
  Percentage of intestinal malrotation among foetuses with abnormal positionning of mesenteric vessels

SECONDARY OUTCOMES:
Rate of correlation between prenatal | day 1
  Rate of correlation between prenatal
Rate of postnatal ultrasound | day 1
  Rate of postnatal ultrasound
type of intestinal malrotation | day 1
  type of intestinal malrotation

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC